CLINICAL TRIAL: NCT06658093
Title: RESTOR [Rapamycin and Everolimus Study Towards Older Rejuvenation]: An Exploratory PK/PD Study of mTOR Inhibition in Older Human Subjects
Brief Title: RESTOR: PK/PD mTORi Inhibition in Older Adults
Acronym: RESTOR
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ellen Kraig, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00000471; U01AG089242 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Aging
Keywords: mTOR inhibitors
MeSH Terms: interventions — Sirolimus; Everolimus

STUDY DESIGN:
Intervention Model Description: A single site open label adaptive clinical trial (Aim 1:Sub-study 2) followed by a placebo-controlled blinded clinical trial (Aim 2) to optimize the use of mTOR inhibitors in older persons a functions of drug, dose, dosing schedule and sex. It will be carried out in 2 sub-studies:
  Aim 1:
  -Sub-study 2: Comparison of 2 mTOR inhibitors in an adaptive open-label dose finding pharmacokinetic/pharmacodynamic study
  Aim 2:
  Sub-study 3: Assess the safety/tolerability/adverse events of optimized dose of mTOR inhibitors in daily vs intermittent dosing
Who Masked: Participant, Care Provider
Masking Description: Blinding will only occur in Aim 2 (Sub-study 3). Randomization will be done by the research pharmacy providing the investigational drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Aim 1:Sub-study 2 Daily dosing Cohort Rapamycin (Experimental): Aim 1 is an open label, adaptive, dose finding PK/PD trial in older women and men.
  In sub-study 2 (part of Aim 1), an older cohort will be studied to determine the optimal dose (OD) in milligrams of rapamycin (RAPA) based on changes in PD parameters 'downstream' from mTOR. Based on the data acquired, additional older cohorts will be tested at higher/lower doses in an adaptive, step-wise trial design.
  Interventions: Drug: Rapamycin
- Aim 1: Sub-study 2 Daily dosing Cohort Everolimus (Experimental): Aim 1 is an open label, adaptive, dose finding PK/PD trial in older women and men.
  In sub-study 2 (part of Aim 1), an older cohort will be studied to determine the optimal dose (OD) of everolimus (EVERO) in milligrams based on changes in PD parameters 'downstream' from mTOR. Based on the data acquired, additional older cohorts will be tested at higher/lower doses in an adaptive, step-wise trial design.
  Interventions: Drug: Everolimus
- Aim 1:Sub-study 2 Intermittent dosing Cohort Rapamycin (Experimental): Aim 1 is an open label, adaptive, dose finding PK/PD trial in older women and men.
  In sub-study 2 (part of Aim 1), an older cohort will be studied to determine the optimal dose (OD) in milligrams and the optimal interval for intermittent delivery of rapamycin (RAPA) based on changes in PD parameters 'downstream' from mTOR. Based on the data acquired, additional older cohorts will be tested at higher/lower doses in an adaptive, step-wise trial design.
  Interventions: Drug: Rapamycin
- Aim 1: Sub-study 2 Intermittent dosing Cohort Everolimus (Experimental): Aim 1 is an open label, adaptive, dose finding PK/PD trial in older women and men.
  In sub-study 2 (part of Aim 1), an older cohort will be studied to determine the optimal dose (OD) in milligrams and the optimal interval for intermittent delivery of everolimus (EVERO) based on changes in PD parameters 'downstream' from mTOR. Based on the data acquired, additional older cohorts will be tested at higher/lower doses in an adaptive, step-wise trial design.
  Interventions: Drug: Everolimus
- Aim 2: Sub-study 3 Optimized DAILY Dose of an mTOR inhibitor (Experimental): Based on the findings from Aim 1, the optimal drug (RAPA or EVERO) and dose for DAILY delivery will be tested in a blinded placebo-controlled trial in older human subjects. The drug/dose used in males may differ from the one used in females as the OD will be determined independently for the two sexes. PD parameters 'downstream' from mTOR will be followed.
  Interventions: Drug: Rapamycin; Drug: Everolimus
- Aim 2: Sub-study 3 Optimized INTERMITTENT Dosing of an mTOR inhibitor (Experimental): Based on the findings from Aim 1, the optimal drug (RAPA or EVERO), interval between doses, and dose for INTERMITTENT delivery will be tested in a blinded placebo-controlled trial in older human subjects. The drug/dose/interval used in males may differ from the one used in females as the OD will be determined independently for the two sexes. PD parameters 'downstream' from mTOR will be followed. Although drug is delivered on an intermittent schedule, subjects will be given a pill each day (either drug or placebo, as scheduled) to maintain blinding.
  Interventions: Drug: Rapamycin; Drug: Everolimus
- Aim 2: Sub-study 3 Placebo control (Placebo Comparator): Daily administration of a placebo will be given to a cohort of older human subjects. Both males and females will be enrolled as controls.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rapamycin — mTOR inhibitor
  Other Names: RAPA
  Arms: Aim 1:Sub-study 2 Daily dosing Cohort Rapamycin; Aim 1:Sub-study 2 Intermittent dosing Cohort Rapamycin; Aim 2: Sub-study 3 Optimized DAILY Dose of an mTOR inhibitor; Aim 2: Sub-study 3 Optimized INTERMITTENT Dosing of an mTOR inhibitor
Drug: Everolimus — mTOR inhibitor
  Other Names: EVERO
  Arms: Aim 1: Sub-study 2 Daily dosing Cohort Everolimus; Aim 1: Sub-study 2 Intermittent dosing Cohort Everolimus; Aim 2: Sub-study 3 Optimized DAILY Dose of an mTOR inhibitor; Aim 2: Sub-study 3 Optimized INTERMITTENT Dosing of an mTOR inhibitor
Other: Placebo — Inert placebo for rapamycin or everolimus
  Other Names: Placebo capsule
  Arms: Aim 2: Sub-study 3 Placebo control

SUMMARY:
As people get older, there are changes in their cells and tissues that may affect their ability to function. This can lead to increased death and age-associated disorders, like heart disease, cancer, and Alzheimer's disease. Studies in animal models have been able to identify drugs that slow the aging process, leading to a longer, healthier life. This study is focused on one such family of drugs, called mTOR inhibitors, and the investigators' goal is to test two of these drugs, Rapamycin (Sirolimus) and Everolimus (Afinitor), in healthy older adults to find a dose and dose timing that can be used to safely inhibit mTOR to the levels seen in young healthy persons. The investigators expect that the dose that works well in women may differ from the one that is best in men, so it is important to include both sexes in this research.

DETAILED DESCRIPTION:
The study will be done in three parts, each with different human subject groups. Participants may only enroll in one of the sub-studies.

Sub-study 1: Determining target mTOR activity values in YOUNG untreated subjects (ages 20-30 years): NOTE: This aim of the study is not a clinical trial, so this population will not be included in participant flow or included as an arm in the study.

This study defines "best dose" as the choice of drug, dose, and frequency that will come closest to restoring the "youthful" levels of mTOR activity in an older individual. The investigators first need to measure mTOR activity in young untreated subjects to define these target "youthful" mTOR activity levels.

Sub-study 2. Finding the most effective drug, dose, and timing for dosing for oral dosing of the mTOR inhibitor drugs in older adults (65-90 years):

Healthy older persons will be recruited for a short-term (6 week treatment plus 4 week follow-up) dose-finding study. The most effective, but safe dose will then be tested in a larger number of subjects in Sub-study 3. Importantly, the best drug and dose regimen for females may differ from the one determined for males so the cohort will include both sexes.

Sub-study 3. Placebo controlled trial testing of DAILY (sustained) vs. INTERMITTENT mTOR inhibition in older human males and females:

Sub-study 3 will enroll healthy older persons (65-90 yrs) for a long-term clinical trial (6 months of treatment plus 6 months of follow-up) with 3 test groups:

i) best DAILY dose/drug; ii) best INTERMITTENT dose/drug/interval, and iii) PLACEBO (a pill that looks identical to the medicine, but has no drug in it).

This study will help find out what effects, good and/or bad, Rapamycin or Everolimus have on older people who take the drug for a longer period of time. The safety of Rapamycin and Everolimus in humans has been tested in prior research studies; however, some side effects may not yet be known in healthy older persons. By completing the entire study, the Research Team hopes to learn more about how older human subjects can best be treated using these drugs (mTOR inhibitors) to help them live longer, healthier lives.

ELIGIBILITY:
Inclusion Criteria:

Older Cohort Sub-study 2 (AIM 1) and Sub-study 3 (AIM 2):

1. Age ≥65 to 90 years
2. Men and women
3. In good health with all medical problems stable.
4. Community-dwelling
5. Agreement to adhere to Lifestyle Considerations throughout study duration.
6. Ability of participant to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Older Cohort Sub-study 2 (AIM 1) and Sub-study 3 (AIM 2):

1. Resident of nursing home or long-term care facility
2. Subjects with diabetes or currently taking glucose lowering medications
3. History of moderate-severe heart disease (New York Heart Classiﬁcation greater than grade II) or pulmonary disease (dyspnea on exertion upon climbing one ﬂight of stairs or less; abnormal breath sounds on auscultation); Moderate to severe valvular heart disease
4. Active cancer or history of cancer treatment within the last 5 years
5. Chronic inﬂammatory condition, autoimmune disease, or infectious processes (e.g., active tuberculosis, HIV, rheumatoid arthritis, systemic lupus erythematosus, acute or chronic hepatitis B or C)
6. History of a coagulopathy or any medical condition requiring anticoagulation (except low dose ASA)
7. Renal insuﬃciency with an estimated glomerular ﬁltration rate of <30ml/min
8. Uncontrolled hypercholesterolemia >350mg/dl or uncontrolled hypertriglyceridemia >500mg/dl
9. Anemia or abnormal blood cell counts: hemoglobin level <9.0g.dl; white blood count <3500/mm3; neutrophil count <2000/ mm3; platelet count <125,000/mm3
10. History of skin ulcers or poor wound healing
11. Active tobacco use (within 6 months)
12. Diagnosis of any disabling neurologic disease such as Parkinson's Disease, Amyotrophic Lateral Sclerosis, multiple sclerosis, cerebrovascular accident with residual deﬁcits (muscle weakness or gait disorder), severe neuropathy, diagnosis of dementia or Clox1 score less than 10 at the time of screening visit, cognitive impairment due to any reason such that the patient is unable to provide informed consent
13. Liver disease
14. Systemic treatment with an immunosuppressant (prednisone, etc.) within the year prior to enrollment
15. Treatment with drugs known to affect cytochrome P450 (CYP3A4), i.e., diltiazem, erythromycin.
16. Patients with history of recent (within 6 months) myocardial infarction or active coronary disease
17. Patients with history of recent (within 6 months) intestinal disorders
18. History of severe head trauma, brain injury, brain surgery, inﬂammation of the brain, or history of seizure disorder
19. History of Long-Covid (PASC) within one year
20. Acute Covid19 or Covid19 infection within the last 6 months
21. Unwilling to forgo grapefruit juice consumption.
22. Participation in mTORi study within the prior year. (Note: participants in AIM 1 will be excluded from participating in AIM 2 of the proposed trial.)
23. Allergic to RAPA or EVERO
24. Allergic to lidocaine
25. Recreational drug use
26. Donated blood over a two-month period prior to study initiation.
27. Currently using cannabidiol (CBD) or tetrahydrocannabinol (THC) or any preparation contained these, or related, substances.
28. Currently using hormone replacement or modulating therapies.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of mTOR inhibitor in blood | Baseline to study end (approximately 12 months for Aim 2; 12 weeks for Aim 1)
  The levels of the study drug will be measured in whole blood
PD measure of inhibition of mTOR activity in blood cells - p-rpS6 | Baseline to study end (approximately 12 months for Aim 2; 12 weeks for Aim 1)
  Proteins prepared from PBMCs (peripheral blood mononuclear cells) will be analyzed for phosphorylation of ribosomal protein S6, downstream of mTORC1.
Level of Soluble Intercellular Adhesion Molecule-1 (sICAM-1) | Baseline to study end (approximately 12 months)
  The level of soluble (s)ICAM-1 will be measured in serum.

SECONDARY OUTCOMES:
PK of mTOR inhibitor in fat (Aim 2 only) | Baseline and study end (approximately 12 months)
  The levels of the study drug will be measure in fat tissue obtained by adipose biopsy
PK of mTOR inhibitor in muscle (Aim 2 only) | Baseline to study end (approximately 12 months)
  The levels of the study drug will be measured in skeletal muscle obtained by biopsy.
PD measure of inhibition of mTOR activity in fat cells (Aim 2 only) - pS6K | Baseline to study end (approximately 12 months)
  Proteins prepared from adipose tissue will be analyzed for phosphorylation of S6kinase, downstream of mTORC1.
PD measure of inhibition of mTOR activity in muscle (Aim 2 only) - pS6K | Baseline to study end (approximately 12 months)
  Proteins prepared from skeletal muscle tissue biopsy will be analyzed for phosphorylation of S6kinase, downstream of mTORC1.
PD measure of inhibition of mTOR activity in PBMCs, S6-kinase | Baseline to study end (approximately 12 months)
  Proteins prepared from PBMCs (peripheral blood mononuclear cells) will be analyzed for phosphorylation of S6kinase, downstream of mTORC1.
PD measure of inhibition of mTOR activity in adipose cells, rpS6 (Aim 2 only) | Baseline to study end (approximately 12 months)
  Proteins prepared from adipose biopsies will be analyzed for phosphorylation of ribosomal protein S6, downstream of mTORC1.
PD measure of inhibition of mTOR activity in muscle rpS6 (Aim 2 only) | Baseline to study end (approximately 12 months)
  Proteins prepared from muscle biopsies will be analyzed for phosphorylation of ribosomal protein S6, downstream of mTORC1.
PD measure of inhibition of mTOR activity in adipose (fat) cells Akt (Aim 2 only) | Baseline to study end (approximately 12 months)
  Proteins prepared from adipose biopsies will be analyzed for phosphorylation of Akt, downstream of mTORC2.
PD measure of inhibition of mTOR activity in muscle Akt (Aim 2 only) | Baseline to study end (approximately 12 months)
  Proteins prepared from muscle biopsies will be analyzed for phosphorylation of Akt, downstream of mTORC2.
PD measure of inhibition of mTOR activity in PBMCs Akt | Baseline to study end (approximately 12 months)
  Proteins prepared from PBMCs will be analyzed for phosphorylation of Akt, downstream of mTORC2.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kraig, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication in a peer review journal

REFERENCES:
- [Background] Kraig E, Linehan LA, Liang H, Romo TQ, Liu Q, Wu Y, Benavides AD, Curiel TJ, Javors MA, Musi N, Chiodo L, Koek W, Gelfond JAL, Kellogg DL Jr. A randomized control trial to establish the feasibility and safety of rapamycin treatment in an older human cohort: Immunological, physical performance, and cognitive effects. Exp Gerontol. 2018 May;105:53-69. doi: 10.1016/j.exger.2017.12.026. Epub 2018 Feb 3. PMID 29408453